CLINICAL TRIAL: NCT02825576
Title: Prevention of Postoperative Events Following Reversal With Sugammadex or Neostigmine
Acronym: P-PERSON
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of Study Personnel
Sponsor: Northern Sydney Anaesthesia Research Institute (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Northern Sydney and Central Coast Area Health Service (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MSD-IIS-54809
Record Dates: First submitted 2016-06-21; First posted 2016-07-07 (Estimated); Last update posted 2023-03-29 (Actual); Status verified 2023-03

CONDITIONS: Pulmonary Complications
MeSH Terms: interventions — Sugammadex; Neostigmine; Glycopyrrolate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sugammadex group (Active Comparator): Sugammadex 2mg/kg intravenously at completion of surgery.
  Interventions: Drug: Sugammadex
- Neostigmine/Glycopyrrolate group (Active Comparator): Neostigmine 50mcg/kg plus Glycopyrrolate 10mcg/kg intravenously at completion of surgery.
  Interventions: Drug: Neostigmine/Glycopyrrolate

INTERVENTIONS:
Drug: Sugammadex — Sugammadex 2mg/kg given for reversal agent
  Other Names: Bridion
  Arms: Sugammadex group
Drug: Neostigmine/Glycopyrrolate — Neostigmine 50 mcg/kg plus Glycopyrrolate 10 mcg/kg given for reversal agent
  Arms: Neostigmine/Glycopyrrolate group

SUMMARY:
The purpose of this study is to determine if the use of sugammadex (compared with neostigmine) reduces the rate of postoperative pulmonary complications (PPCs).

DETAILED DESCRIPTION:
This is a local, multi-centre, prospective, randomised, double blinded trial of 976 patients.

Objectives:

The primary objective is to determine if the use of sugammadex (compared with neostigmine) reduces the rate of postoperative pulmonary complications (PPCs). Secondary objectives are to determine if the use of sugammadex compared with traditional reversal agents improves patient quality of recovery, reduces the rate of postoperative nausea and vomiting and reduces the rate of airway complications in the Post Anaesthesia Care Unit (PACU).

Study procedures:

Following informed consent prior to surgery, patients will be randomised to two groups allocating drugs used for reversal of muscle relaxation;

1. 2mg/kg sugammadex
2. 50mcg/kg neostigmine with 10mcg/kg glycopyrrolate

Randomisation will be via computer generated numbers, which will be sealed in opaque, sequentially numbered envelopes.

Treating anaesthetist and staff assessing outcomes will be blinded to treatment.

Patients will have neuromuscular transmission (NMT) monitoring intraoperatively to ensure return of train-of-four count (TOFC) >2 prior to reversal. Muscle relaxant will be limited to rocuronium or vecuronium, at the choice of the individual anaesthetist. As this study is planned to be a 'real world' trial, mode of anaesthesia, analgesia, postoperative nausea and vomiting (PONV) prophylaxis and time of reversal will be determined by the individual treating anaesthetist.

Postoperative outcome data will be collected in the recovery unit, on postoperative day 1 and 2 (if still an inpatient), at hospital discharge and via a 30 day post-operative phone call.

Statistical Analysis:

Conservatively estimating the baseline incidence of PPC at 7% baseline incidence and an equally conservative estimate that sugammadex can reduce this to 3% would produce a clinically relevant number needed to treat (NNT) of 29. Accepting an alpha error of 0.05 and beta error of 0.2 would require 930 patients. Allowing for 5% incomplete data and loss to follow up requires 976 patients.

Groups will be analysed on an intention-to-treat basis

1. PPC rate, QoR-15 score and hospital stay will be assessed as continuous variables
2. Post operative Nausea and Vomiting (PONV) score will be assessed as an ordinal variable
3. Mortality and the presence of respiratory and PACU events will be assessed as categorical variables.

The effect of sugammadex on continuous variables will be analysed by 2-tailed Student T-test. The effect of sugammadex on ordinal and categorical variables will be analysed by Chi-squared tests. Binomial regression analysis will be performed on the categorical outcomes for the subgroup analyses. Logistic regression will be performed to analyse the effect of PONV risk on PONV scores.

Appropriate statistical tests to confirm test assumptions are met will be performed. In the case of non-parametric data, the appropriate test will be performed. Interim analysis is planned after 50% data completion.

ELIGIBILITY:
Inclusion Criteria:

* age >18
* patients presenting for non-cardiac surgery
* planned operative time of over 1 hour
* plan to be intubated and to receive muscle relaxants for their surgery
* plan to stay at least one night in hospital

Exclusion Criteria:

* Previous recruitment to the trial
* Hypersensitivity to any of the study drugs
* Patient refusal
* Cognitive Impairment, or language proficiency leading to inability to complete QoR-15 questionnaire
* Body Mass Index (BMI) >40
* Planned postoperative intubation and ventilation
* Liver failure with Child-Pugh class B/C
* Renal failure with either regular peritoneal or haemodialysis or serum creatinine >140mcgmol/L
* Women lactating, pregnant or of childbearing potential who are not willing to avoid pregnancy during the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-12-03 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Incidence of post operative pulmonary complications. | Up to day 2 post operatively.
  Incidence of Postoperative pulmonary complications as defined by The Assess Respiratory Risk in Surgical Patients in Catalonia (ARISCAT) group.

SECONDARY OUTCOMES:
Quality of Recovery Score (QoR-15) | Day 1 and Day 30 post operatively
  A 15- item patient-rated post operative questionnaire designed to assess the early postoperative health status of patients after anesthesia and surgery.
Incidence of post operative nausea and vomiting. | Day of surgery.
  Post Operative Nausea and Vomiting (PONV) Score:
  1. - no PONV
  2. - PONV responsive to antiemetics
  3. - PONV unresponsive to antiemetics
Incidence of airway events in the Post Anaesthesia Care Unit (PACU). | Day of surgery.
  Proportion of patient that exhibit one or more of the following PACU Events (recorded by recovery room nursing staff);
  1. Any desaturation to oxygen saturation by pulse oximetry (SpO2) <90%
  2. Need for manual airway support
  3. Need for oropharyngeal or nasopharyngeal airway
  4. Need for reintubation in PACU
  5. Need for anaesthetist to review the patient
  6. Unplanned Intensive Care Unit (ICU) admission
Mortality | 30 day
  Death of patient within time frame.
Hospital stay | 30 days
  Duration of hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Ben L Olesnicky, BMBS BSc, Principal Investigator — Northern Sydney Anaesthesia Research Institute
Locations (1):
- Royal North Shore Hospital, St Leonards, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Olesnicky B, Doane M, Farrell C, Knoblanche G, Delaney A. Prevention of Postoperative Events following Reversal with Sugammadex or Neostigmine (the P-PERSoN Trial): Pilot Data Following Early Termination of a Prospective, Blinded, Randomised Trial. Anesthesiol Res Pract. 2022 Jul 8;2022:4659795. doi: 10.1155/2022/4659795. eCollection 2022. PMID 35844810